CLINICAL TRIAL: NCT06270953
Title: Impact of Non-invasive Continuous Patient Monitoring System on Patient Management and Health Outcomes
Brief Title: Non-invasive Monitoring: Impact on Patient Management and Outcomes
Status: Completed | Type: Observational
Sponsor: Turtle Shell Technologies Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: DZ_NX_US
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2024-02

CONDITIONS: No Specific Medical Conditions or Disease States

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Obervational group: Patients admitted in the SNF facility during the study period
  Interventions: Device: Dozee Pro NX
- Control group: Historical control with patients admitted in the SNF before the study period

INTERVENTIONS:
Device: Dozee Pro NX — Dozee Pro NX to measure Heart Rate, Respiratory Rate, SPO2 and movements
  Groups: Obervational group

SUMMARY:
Enhancing patient monitoring in SNFs and ALFs is crucial due to challenges in recognizing deteriorating health. Gaps in vital sign checks lead to missed indicators and adverse outcomes. Turtle Shell Technologies' Dozee Pro NX offers continuous non-invasive monitoring, alerting healthcare providers of vital sign changes. This clinical study aims to evaluate Dozee Pro Nx's impact on patient outcomes, practitioner efficiency, and healthcare costs in SNFs and ALFs, addressing gaps in care delivery.

DETAILED DESCRIPTION:
In skilled nursing facilities (SNFs) and assisted living facilities (ALFs), managing patient health presents considerable hurdles in accurately identifying and responding to deteriorating conditions. The intricacies of care within these settings are compounded by a high patient-to-healthcare provider ratio, often leading to infrequent vital sign checks with significant time gaps between assessments. This monitoring gap may result in overlooking early signs of health decline, potentially causing adverse patient outcomes. A February 2014 report by the Office of Inspector General (OIG) underscored this issue, revealing that around 22% of Medicare beneficiaries experienced adverse events during their stays in SNFs, with an additional 11% facing temporary harm events. Notably, 59% of these incidents were considered preventable, largely due to insufficient patient monitoring, care delays, and substandard treatment. In response to these challenges, Turtle Shell Technologies (TST) Private Limited has developed Dozee Pro NX, an innovative system tailored to improve patient monitoring in these healthcare settings. This system employs non-invasive sensors to continuously monitor crucial parameters such as heart rate, respiration rate, blood pressure, temperature, and SpO2. Distinguished from traditional patient monitoring devices, Dozee Pro Nx offers advanced functionalities, including customizable notifications to alert healthcare providers of vital sign deterioration, thereby enabling prompt intervention. The primary objective of this clinical study is to evaluate the potential impact of the Dozee Pro Nx system on patient outcomes, healthcare practitioner efficiency, and overall healthcare costs. This investigation aims to ascertain whether the implementation of this advanced monitoring technology can effectively address the identified gaps in patient care within SNFs and ALFs, ultimately leading to improved health outcomes and enhanced care delivery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Weight between 40kg-120kgs

Exclusion Criteria:

* Terminal illness with a life expectancy of less than 1 month.
* Have any condition that could interfere with the subject's ability to lie flat or stable on the bed
* Needs the use of equipment whose operation can interfere with Investigation System operations
* Patients planned to be transferred from the facility within 72 hours
* Prisoners
* Pregnant

Ages: 18 Months to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted on subjects in the age group above 18 years regardless of gender. The study is done on patients admitted in the SNF who fulfill the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Care Escalation and/or Transfers (Subgroup- ER visits, Surgical Interventions & Hospitalizations, ICU Admissions), | 3 months

SECONDARY OUTCOMES:
HCP experience response data | 3 Months
Care pathway mapping | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Darthard, LNFA, Principal Investigator — Oak Village Healthcare
Locations (1):
- Oak Village Healthcare, Lake Jackson, Texas, United States

IPD SHARING:
Plan to Share IPD: No